CLINICAL TRIAL: NCT01699828
Title: Exploring Occupancy of Dopamine D3 Receptor by Buspirone in Humans Using PET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, PI, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 186/2011
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Smoking Cessation; Tobacco Use Cessation
Keywords: buspirone; smoking cessation; dopamine; PET imaging; [11C]-(+)-PHNO
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation | interventions — Buspirone; Lactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Buspirone 120 mg (Experimental): Buspirone 120 mg (encapsulated).
  Interventions: Drug: Buspirone
- Buspirone 60 mg (Experimental): Buspirone 60 mg (encapsulated)
  Interventions: Drug: Buspirone
- Placebo (Placebo Comparator): Placebo (encapsulated)
  Interventions: Drug: Placebo
- Buspirone 30 mg (Experimental): Buspirone 30 mg (encapsulated).
  Interventions: Drug: Buspirone

INTERVENTIONS:
Drug: Buspirone — The buspirone will be given once as a tablet and encapsulated for blinding.
  Other Names: Buspar
  Arms: Buspirone 120 mg; Buspirone 30 mg; Buspirone 60 mg
Drug: Placebo — Placebo will be lactose and encapsulated for blinding. A single capsule will be given.
  Other Names: lactose
  Arms: Placebo

SUMMARY:
The objective of the present study is to use positron emission tomography brain imaging to investigate D3 occupancy of buspirone, an FDA-approved anxiolytic which acts as a serotonin partial agonist but has recently been identified as a D3 antagonist. It is hypothesized that clinically relevant doses of buspirone will occupy the D3 receptor.

DETAILED DESCRIPTION:
Buspirone is used for anxiety disorder treatment, a therapeutic effect that has been thought to be mediated through its partial agonist properties at the serotonin receptor. However, since one PET study in humans has shown low occupancy of the serotonin by buspirone in clinical doses and since the DRD3 has been recently implicated in anxiety, some therapeutic effects of buspirone may be mediated through the DRD3. In human clinical studies, promising effects of buspirone have been reported for treatment of substance dependence, including tobacco, marijuana, and opiates, and clinical studies in cocaine dependent subjects are underway. However, it is unclear if buspirone is producing those effects through the DRD3 and no human study has incorporated a PET imaging component to investigate this question; it remains unclear whether buspirone significantly occupies the DRD3 at therapeutic doses in humans.

ELIGIBILITY:
Inclusion Criteria:

- 19 years or older

Exclusion Criteria:

* Medical condition including cardiovascular, renal, hepatic or cerebrovascular diseases
* History of or current neurological illnesses including seizure disorders, migraine, multiple sclerosis, movement disorders, head trauma, CVA or CNS tumor, - Present or past psychiatric condition including mood, anxiety, psychotic disorders and substance abuse and/or dependence.
* Condition that precludes use of buspirone or that will interfere with participation in the present study (such as hypersensitive to buspirone hydrochloride).
* Pregnancy or breastfeeding.
* Presence of metal objects in the body or implanted electronic devices, that preclude safe MR scanning.
* Claustrophobia.
* Current use or use during the previous month of medication that may affect the CNS, including monoamine oxidase inhibitor (MAOI) or positive during drug screening for drugs of abuse or any medication that could increase the risk of buspirone administration.
* Exposure to radiation in the last 12 month exceeding permissible limit for subjects participating in research.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Dose-response occupancy of buspirone at DRD3 | few months
  [11C]-(+)-PHNO binding potential at three doses of buspirone and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Boileau, PhD, Principal Investigator — Center for Addiction and Mental Health; Bernard Le Foll, MD, PhD, Principal Investigator — Center for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.net/research